CLINICAL TRIAL: NCT06158217
Title: Effect of Ultrasound Combined With Microbubbles on Blood Perfusion in Invasive Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MR-11-22-009539
Record Dates: First submitted 2023-11-09; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-06

CONDITIONS: Invasive Breast Cancer; Cavitation; Perfusion
Keywords: Contrast-enhanced ultrasound; ultrasound combined with microbubbles; Invasive ductal carcinoma of breast
MeSH Terms: conditions — Carcinoma, Ductal, Breast | interventions — Microbubbles

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: ultrasound combined with microbubbles — IBC tumors were treated with microbubbles (MBs) stimulated by ultrasound
  Other Names: Cavitation effect; Microbubble assisted ultrasound technique

SUMMARY:
Blood perfusion insufficiency and hypoxia are the main causes of drug resistance to chemotherapy in breast cancer. Increasing blood perfusion can improve drug delivery. The cavitation effect of ultrasound-stimulated microbubbles (USMBs) is known to enhance tumor blood perfusion, so we conducted a prospective human study to investigate the effects of USMBs on hemoperfusion in invasive breast cancer (IBC).

DETAILED DESCRIPTION:
patients with IBC were selected from the breast surgery department of our hospital. To induce an enhanced perfusion effect, IBC tumors were treated with SonoVue® microbubbles (MBs) stimulated by ultrasound, with a mechanical index (MI) of 0.2-0.3; 1 mL of SonoVue® MBs were injected at 3.5-min intervals three times for a USMB treatment lasting 10 min. The contrast-enhanced ultrasound (CEUS) parameters peak intensity (PI), area under the curve (AUC), and perfusion area were used to evaluate the changes in blood perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Invasive Breast Cancer
* patients scheduled to undergo surgical resection
* maximum lesion diameter < 4 cm
* age over 18 years

Exclusion Criteria:

* patients with allergies to SonoVue®
* patients with severe cardiopulmonary insufficiency,
* patients who had already received neoadjuvant chemotherapy
* pregnant women
* individuals with mental illness
* Patients who refused to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Invasive breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2025-05-06 (Estimated); Study Completion 2025-05-06 (Estimated)

PRIMARY OUTCOMES:
changes in peak intensity (PI) | 15 minutes after the USMB procedure
  PI represents the quantitative scale of the highest average concentration of microbubble (MB) in the region of interest (ROI); thus, a larger PI corresponds to a higher concentration of MB in the ROI.
area under the curve (AUC) | 15 minutes after the USMB procedure
  AUC represents the total amount of MB passing through the ROI during perfusion; thus, a larger AUC corresponds to greater perfusion in the ROI.
percentage increase in the perfusion area (%) of tumor | 15 minutes after the USMB procedure
  The percentage increase in the perfusion area (%) was calculated as follows: (perfusion area after the USMB procedure - perfusion area before the USMB procedure) × 100%/perfusion area before the USMB procedure. The greater "percentage increase of perfusion area (%)", the more significant the improvement of blood perfusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Dong Y, Zhang D, Feng W, Huang Y, Ge Z, Shi XQ. Effect of Ultrasound Combined with Microbubbles on Blood Perfusion in Invasive Breast Cancer-A Prospective Clinical Trial. Technol Cancer Res Treat. 2026 Jan-Dec;25:15330338261423051. doi: 10.1177/15330338261423051. Epub 2026 Feb 8. PMID 41656585